CLINICAL TRIAL: NCT03178773
Title: Trial to EXamine Text Messaging for Diabetes in ED Patients Incorporating Social Support - Intervention With Washout
Brief Title: TExT-MED + FANS Full Trial
Acronym: TExTMED+FANSII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Elizabeth Burner, Assistant Professor of Clinical Emergency Medicine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-17-00406
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Results first posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Diabetes
Keywords: mobile health; social support; health disparity; Latino
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TExT-MED only (Active Comparator): Patients receive SMS-textmessage curriculum to improve self0-efficacy and self care for diabetes. A patient-identified family member receives a social support curriculum (FANS) in traditional booklet form.
  Interventions: Behavioral: TExT-MED
- TExT-MED+FANS (Experimental): Patients receive SMS-textmessage curriculum to improve self0-efficacy and self care for diabetes. A patient-identified family member receives a social support curriculum (FANS) by SMS-text-message synchronized by time and content.
  Interventions: Behavioral: TExT-MED; Behavioral: FANS

INTERVENTIONS:
Behavioral: TExT-MED — messages designed to inspire motivation and behavior change
Behavioral: FANS — SMS delivered messages to family members to improve social support
  Arms: TExT-MED+FANS

SUMMARY:
This is an intervention to study incorporating social support into mHealth interventions for low-income, ED patients with diabetes

DETAILED DESCRIPTION:
Diabetes has disproportionately affected the Latino population. TExT-MED (Trial to Examine Text Message for Emergency Department Patients with Diabetes) is a locally designed, successful mobile health (mHealth) intervention for low income Latinos with diabetes. Social support interventions have likewise been successful at improving patient self-efficacy and disease management but are limited in scale due to two key obstacles: 1) requirements of in-person training of family and friends to be supporters and 2) the need to coordinate schedules and physical location between the patient and their supporter. mHealth can overcome these obstacles by allowing supporters to be trained remotely via a mobile platform and by allowing communication between a patient and supporter to occur at any time or place. The proposed intervention leverages the success of TExT-MED by augmenting the program with a social supporter that each patient can select from his or her own social support system (Family And friend Network Supporters (FANS)), creating TExT-MED+FANS. This is a 12 month, randomized study of this intervention. At the completion of the trial, we will evaluate the user experience with TExT-MED+FANS, and the impact of TExT-MED+FANS on patient motivation, self-efficacy and behaviors through a qualitative analysis of semi-structured individual interviews.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* HbA1c>8.5
* Social support person identified and contacted

Exclusion Criteria:

* unable to consent
* does not speak/read English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- LAC+USC Medicine Center Emergency Department, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burner E, Hazime D, Menchine M, Mack W, Mercado J, Aleman A, Hernandez Saenz A, Arora S, Wu S. mHealth Social Support Versus Standard Support for Diabetes Management in Safety-Net Emergency Department Patients: Randomized Phase-III Trial. JMIR Diabetes. 2025 Apr 23;10:e56934. doi: 10.2196/56934. PMID 40266665

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TExT-MED Only | TExT-MED+FANS
Started | 86 | 80
3month Phone Follow up | 49 | 51
6month in Person Follow up | 54 | 46
9month Follow up Phone | 36 | 51
Completed | 47 | 40
Not Completed | 39 | 40
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 29 | 25
Not completed — Withdrawal by Subject | 10 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 86 | 80 | 166
Age, Continuous [Mean (Inter-Quartile Range); unit: years] — Age: collected from medical records
  years | 50.7 [40.7 to 55.4] | 47.7 [41.6 to 53.4] | 48.9 [40.7 to 55.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 35 | 84
  Male | 37 | 45 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity: Collected by patient self-report, with option for decline to state
  Participants
    Hispanic or Latino | 82 | 74 | 156
    Not Hispanic or Latino | 3 | 6 | 9
    Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race: collected by patient self-report, with option for more than one race and decline to state
  Participants
    American Indian or Alaska Native | 2 | 3 | 5
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 6 | 9
    White | 40 | 34 | 74
    More than one race | 2 | 1 | 3
    Unknown or Not Reported | 37 | 36 | 73
Region of Enrollment [Number; unit: participants]
  United States | 86 | 80 | 166
Language Preferred [Count of Participants; unit: Participants]
  Spanish | 64 | 52 | 116
  English | 22 | 28 | 50
Born outside US [Count of Participants; unit: Participants] | 75 | 56 | 131
HbA1c [Median (Inter-Quartile Range); unit: % percentage of hemoglobin glycosylated] | 10.3 [9.70 to 12.0] | 10.6 [9.60 to 12.0] | 10.4 [9.70 to 12.0]
BMI [Mean (Standard Deviation); unit: kg^m2] — BMI: calculated from Weight and Height. As a measure of adiposity, it correlates positively with cardiovascular disease outcomes. While imperfect, it is an easily measured and validated marker. Population: 2 participants were unable to stand to provide height
  kg^m2
    number analyzed (Participants) | 84 | 80 | 164
    (all) | 30.78 (7.96) | 29.34 (7.18) | 30.07 (7.60)
Abdominal circumference (cm) [Mean (Standard Deviation); unit: cm] — A measure of central adiposity, it correlates with cardiovascular outcomes. Population: 20 participants were unable to provide abdominal circumference measurement
  cm
    number analyzed (Participants) | 78 | 68 | 146
    (all) | 138.67 (174.29) | 104.82 (16.61) | 122.90 (128.63)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Systolic blood pressure mmHg: Blood pressure is measured by study RAs after the patient is seated for 5 minutes, with the average of three readings used as the systolic blood pressure for that visit. Systolic blood pressure is associated with cardiovascular complications
  mmHg | 131.55 (25.02) | 131.03 (28.90) | 131.30 (26.88)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure is measured by study RAs after the patient is seated for 5 minutes, with the average of three readings used as the diastolic blood pressure for that visit.
  mmHg | 79.98 (15.81) | 81.61 (16.15) | 80.77 (15.95)
Summary of Diabetes Self-Care Activities [Mean (Standard Deviation); unit: units on a scale] — Summary of Diabetes Self-care Activities (Toobert, Hampson, Glasgow, & RE, 2000). The Summary consists of 6 subscales representing different domains of diabetes related healthy behaviors and self-care. It has been validated in over 10 studies, with the results published in two manuscripts: one with three studies (Toobert & Glasgow, 1994), and one with seven studies(Toobert et al., 2000). Each measure ranges from Each range from 0-7, indicating number of days per week patient reports engaging in these behaviors.
  units on a scale
    Following a generally healthy diet | 3.38 (2.44) | 3.07 (2.51) | 3.23 (2.47)
    Following a disease specific diet plan | 3.98 (1.90) | 3.74 (1.89) | 3.87 (1.90)
    Self-monitoring blood glucose as advised by a h | 2.55 (2.79) | 2.76 (3.06) | 2.65 (2.92)
    Checking feet daily for wounds | 4.01 (3.00) | 4.11 (2.86) | 4.06 (2.93)
    Spacing carbohydrates throughout the day | 2.78 (2.65) | 3.00 (2.46) | 2.89 (2.56)
    Getting sufficient physical activity | 2.51 (2.62) | 2.43 (2.53) | 2.47 (2.57)
Wilson 3 Item Scale [Mean (Standard Deviation); unit: units on a scale] — Medication adherence(Wilson et al.,2014). The 3item medication adherence scale is a self-report measure that assessing no. of days medication missed in prior month, days taken medication as advised & self-rated medication adherence. Developed in HIV research, it has been validated for non-HIV medications (Wilson, et al,2016). Each component contributes 33% of the scale. Total score ranges from 0-100. It is the combination of 3 sub-scores, (days missed dose(negative scored), self-rating, days taking medications as indicated). Higher scores indicate better medication adherence. Population: 1 participant decline to answer questions
  units on a scale
    number analyzed (Participants) | 85 | 80 | 165
    (all) | 67.16 (31.13) | 65.85 (28.23) | 66.53 (29.67)
Healthcare Utilization [Mean (Standard Deviation); unit: Number of Healthcare Encounters] — Healthcare utilization by the patients' report of clinic appointments, ED visits and hospitalizations within enrollment through 6 months at each follow up visit. EMR review used instead, as self-report was inconsistent.
  Number of Healthcare Encounters
    ED/UCC Visits | 2.45 (2.12) | 2.38 (3.29) | 2.42 (2.74)
    Hospitalization | 0.43 (0.80) | 0.44 (0.78) | 0.43 (0.79)
    Clinic Visits Made | 3.28 (5.61) | 2.74 (5.25) | 3.02 (5.43)
Diabetes Empowerment Scale Short Form [Mean (Standard Deviation); unit: units on a scale] — Self-efficacy (Diabetes Empowerment Scale Short Form) (Anderson, Fitzgerald, Gruppen, Funnell, & Oh, 2003), is a measure of a patient's overall diabetes related self-efficacy, shortened by the original from 37 to an 8 item scale. It has reliability of alpha=0.84; and has been shown to be sensitive to change in multiple populations and is correlated with improved glycemic control measured by A1C (Anderson et al., 2003). It ranges from 8-40 points; higher score indicates higher self-efficacy.
  units on a scale | 30.50 (5.56) | 31.09 (4.99) | 30.78 (5.28)
Diabetes Distress Scale [Mean (Standard Deviation); unit: units on a scale] — (Diabetes Distress Scale) (Polonsky et al., 2005), is a 17 item scale measuring distress related to emotional burden, physician-related distress, regimen-related distress, and diabetes-related interpersonal issues. It has a Cronbach's alpha of 0.88-0.93 in various studies. Higher scores are negatively correlated with several healthy behaviors. Each question is a Likert scale ranking of how serious a particular issue is from 1-6, 6 indicating a more significant problem. The scores are then averaged across all item, with final scores ranging from 1-6, with 6 indicating higher levels of distress. Population: 11 participants decline to answer questions
  units on a scale
    number analyzed (Participants) | 80 | 75 | 155
    (all) | 2.32 (0.86) | 2.60 (1.11) | 2.46 (0.10)
Patient Health Questionnaire 9 [Mean (Standard Deviation); unit: units on a scale] — Depression as measured by the PHQ-9 (Kroenke, Spitzer, Williams, & Lowe, 2010), is a widely used scale of depression used in clinical practice and research. The Cronbach's alpha ranges from 0.86-0.89, and it has been validated in multiple languages. Depression is worse with higher scores. Score ranges from 0 to 27. Higher levels of depression are associated with fewer healthy behaviors and worse glycemic control.
  units on a scale | 8.90 (6.94) | 9.45 (6.31) | 9.16 (6.63)
Fatalism [Mean (Standard Deviation); unit: units on a scale] — Fatalism is measured by the Diabetes Fatalism Scale (Egede & Ellis, 2010), which measures three subscale emotional distress, religiosity and coping and perceived self-efficacy, which are summed together. The total score ranges from 12-72, higher score indicates higher fatalism, and has a Cronbach's alpha of 0.80. The score is associated with glycemic control, depression, self-care behaviors and social factors.
  units on a scale | 34.09 (9.90) | 35.86 (9.85) | 34.94 (9.89)
WHO Quality of life [Mean (Standard Deviation); unit: units on a scale] — Quality of life (World Health Organization WHO-5 Well Being Index) (Topp, Ostergaard, Sondergaard, & Bech, 2015) is a widely used measure of quality life, validated in many languages and consists of only 5 items. Each self-reported item is scored between 0 and 5, summed together and then multiplied by 4. The total range is from 0 to 100, with 0 being the lowest quality of life.
  units on a scale | 61.91 (26.59) | 58.00 (29.48) | 60.02 (28.00)
Diabetes Family Behavior Checklist [Mean (Standard Deviation); unit: units on a scale] — Diabetes-related supportive and obstructive family behaviors are measured by patient report on the Diabetes Family Behavior checklist (Lewin et al., 2005). Family behaviors: supportive and non-supportive sub-scores of the Diabetes Family Behavior Checklist: supportive ranges from 4-45 (4 being lowest in family supportive behavior), non-supportive ranges from 7-35 (4 indicating least report of non-supportive behavior). Non-supportive scores are subtracted form supportive scores for a total.
  units on a scale
    Supportive | 23.65 (9.12) | 24.56 (9.32) | 24.09 (9.20)
    Non-Supportive | 18.27 (7.23) | 19.28 (7.22) | 18.75 (7.22)
Diabetes Care Profile Support [Mean (Standard Deviation); unit: units on a scale] — Diabetes-specific social support is measured by the Diabetes Care Profile Support Questions,(Fitzgerald et al., 1996) with sub-scores for perceived disease specific support needs and perceived disease specific support received. Diabetes Care Profile support questions: Support wanted, and support received. Each range from 5 to 30, high scores indicating high desire for support and higher support received.
  units on a scale
    Perceived Disease Specific Support Needs | 23.22 (7.51) | 24.04 (7.55) | 23.61 (7.52)
    Perceived Disease Specific Support Received | 17.91 (8.81) | 19.16 (9.06) | 18.51 (8.92)
    Support Attitudes | 6.58 (5.50) | 6.39 (4.68) | 6.49 (5.11)
Norbeck Social Support Questionnaire [Mean (Standard Deviation); unit: units on a scale] — General social support is captured by the Norbeck Social Support Questionnaire Emotional and&Tangible subscales.(Norbeck, Lindsey, & Carrieri, 1981) General social support: Norbeck Social Support Questionnaire, emotional sub score (ranges 0-16, with higher scores indicating higher perceived emotional support) & tangible sub score (0-8, higher score indicating higher perceived tangible support). While the subscores are highly correlated, the authors do not recommend Cronbach's alpha as a test of internal validity.(http://eileengigliotti.com/uploads/1/1/0/2/110241155/nssq-psychometric.pdf) Population: 14 participants decline to answer questions
  units on a scale
    Emotional: number analyzed (Participants) | 77 | 75 | 152
    Emotional | 14.00 (3.32) | 13.68 (3.15) | 13.84 (3.23)
    Tangible: number analyzed (Participants) | 77 | 75 | 152
    Tangible | 6.83 (1.77) | 7.15 (1.57) | 6.99 (1.68)
Partner Distress Scale - Total [Mean (Standard Deviation); unit: units on a scale] — Supporter diabetes-related distress is measured by the Partner Distress Scale (Polonsky, Fisher, Hessler, &Johnson, 2016). The self-report scale consists of 21 items in 4 domains: "my partner's diabetes management", "how best to help", "diabetes & me", & "hypoglycemia". Domains are summed together. Each item is score from 0 to 4, lower scores indicate less distress. The total score is an average of the 21 items. The Cronbach's alpha was 0.76 for total scores. Greater partner distress is correlated with higher A1C among patients, worse self-care & lower satisfaction with relationship Population: 1 participant decline to answer question
  units on a scale
    number analyzed (Participants) | 85 | 80 | 165
    (all) | 1.32 (0.94) | 1.52 (0.95) | 1.42 (0.95)

OUTCOME MEASURES:

1. Primary Outcome: Change in HBA1c From Baseline
Description: Glycemic control is measured by hemoglobin A1C collected at point-of-care from an Afinion AS100 capillary point of care machine. The Afinion machine has excellent point of care correlation with laboratory values. As a surrogate for average glycemic control over the previous 3 months and with correlation with clinical outcomes, hemoglobin A1c is a marker of overall clinical disease management. Change is baseline value minus follow up value.
Time Frame: 6 Months
Population: 2 of the HbA1c were collected from electronic healthcare records in the active control group. 1 intervention group patient refused blood draw at follow up.
Measure: Mean (95% Confidence Interval); unit: %mmHg/dL
Arm/Group | TExT-MED Only | TExT-MED+FANS
Number analyzed (Participants) | 54 | 45
%mmHg/dL | 1.42 [.83 to 2.02] | 1.34 [.53 to 2.15]

2. Secondary Outcome: Change in HBA1c From 6 Months to 12 Months
Description: Glycemic control is measured by hemoglobin A1C collected at point-of-care from an Afinion AS100 capillary point of care machine. The Afinion machine has excellent point of care correlation with laboratory values. As a surrogate for average glycemic control over the previous 3 months and with correlation with clinical outcomes, hemoglobin A1c is a marker of overall clinical disease management. Change is 6 month value minus 12 month value.
Time Frame: 12 months
Population: 2 intervention group patient refused blood draw at follow up.
Measure: Mean (95% Confidence Interval); unit: %mmHg/dL
Arm/Group | TExT-MED Only | TExT-MED+FANS
Number analyzed (Participants) | 47 | 38
%mmHg/dL | -.36 [-.93 to .22] | .28 [-.30 to .86]

3. Secondary Outcome: Change in BMI From Baseline
Description: Calculated from Weight and Height. As a measure of adiposity, it correlates positively with cardiovascular disease outcomes. While imperfect, it is an easily measured and validated marker.
Time Frame: 6 Months
Population: 4 participants were not able to stand on the scale to measure weight
Measure: Mean (Standard Deviation); unit: kg^m2
Groups:
- Total: Both arms combined
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 50 | 46 | 96
kg^m2 | -7.91 (33.80) | -3.84 (22.94) | -5.96 (29.03)

4. Secondary Outcome: Change in BMI From 6 Months to 12 Months
Description: as for outcome 3
Time Frame: 12 Months
Population: 5 participants unable stand to provide weight
Measure: Mean (Standard Deviation); unit: kg^m2
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 45 | 37 | 82
kg^m2 | -3.38 (22.51) | 4.02 (24.88) | -0.04 (23.75)

5. Secondary Outcome: Change in Abdominal Circumference From Baseline
Description: A measure of central adiposity, it correlates with cardiovascular outcomes.
Time Frame: 6 Months
Population: abdominal circumference unable to be collected from 20 patients
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 43 | 37 | 80
cm | 1.58 (14.70) | 2.73 (22.54) | 2.11 (18.62)

6. Secondary Outcome: Change From Abdominal Circumference From 6 Months to 12 Months
Description: A measure of central adiposity, it correlates with cardiovascular outcomes.
Time Frame: 12 Months
Population: abdominal circumference not measured in 9 participants
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 44 | 34 | 78
cm | 0.99 (5.10) | 0.85 (18.51) | 0.93 (12.70)

7. Secondary Outcome: Change in Systolic Blood Pressure From Baseline
Description: Blood pressure is measured by study RAs after the patient is seated for 5 minutes, with the average of three readings used as the systolic blood pressure for that visit. Systolic blood pressure is associated with cardiovascular complications
Time Frame: 6 Months
Population: 2 participants in active control arm did not attend follow up visit. Hba1c taken from medical records, no other data available. 2 participants refused BP measurement
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 50 | 46 | 96
mmHg | -9.11 (30.45) | -13.07 (36.34) | -11.00 (33.28)

8. Secondary Outcome: Change in Systolic Blood Pressure From 6 Months to 12 Months
Description: as for outcome 7
Time Frame: 12 Months
Population: 11 patients with SBP unable to be obtained
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 41 | 35 | 76
mmHg | -4.95 (31.81) | 2.09 (37.46) | -1.71 (34.47)

9. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline
Description: Blood pressure is measured by study RAs after the patient is seated for 5 minutes, with the average of three readings used as the diastolic blood pressure for that visit.
Time Frame: 6 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 50 | 46 | 96
mmHg | -0.27 (17.11) | -2.56 (20.09) | -1.36 (18.53)

10. Secondary Outcome: Change in Diastolic Blood Pressure From 6 Months to 12 Months
Description: as for outcome 9
Time Frame: 12 Months
Population: 11 patients with DBP unable to be obtained
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 41 | 35 | 76
mmHg | -0.82 (17.39) | 5.20 (20.15) | 1.95 (18.82)

11. Secondary Outcome: Change in Summary of Diabetes Self-care Activities From Baseline
Description: Summary of Diabetes Self-care Activities (Toobert, Hampson, Glasgow, & RE, 2000). The Summary consists of 6 subscales representing different domains of diabetes related healthy behaviors and self-care. It has been validated in over 10 studies, with the results published in two manuscripts: one with three studies (Toobert & Glasgow, 1994), and one with seven studies(Toobert et al., 2000). Each measure ranges from Each range from 0-7, indicating number of days per week patient reports engaging in these behaviors.
Time Frame: 6 Months
Population: 2 participants in active control arm did not attend follow up visit. Hba1c taken from medical records, no other data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 52 | 46 | 98
units on a scale
  Following a generally healthy diet | -1.55 (2.91) | -1.17 (2.69) | -1.37 (2.80)
  Following a disease specific diet plan | -0.42 (2.12) | -0.78 (1.93) | -0.59 (2.03)
  Self-monitoring blood glucose as advised by a h | -0.91 (3.00) | -0.10 (2.84) | -0.53 (2.94)
  Checking feet daily for wounds | -1.25 (2.96) | -1.36 (2.69) | -1.30 (2.83)
  Spacing carbohydrates throughout the day: number analyzed (Participants) | 52 | 45 | 97
  Spacing carbohydrates throughout the day | -0.71 (4.34) | -0.20 (3.31) | -0.47 (3.89)
  Getting sufficient physical activity | -0.39 (2.99) | -0.90 (3.14) | -0.63 (3.06)

12. Secondary Outcome: Change in Summary of Diabetes Self-care Activities From 6 Months to 12 Months
Description: as for outcome 11
Time Frame: 12 Months
Population: one participant did not answer carb spacing as they did not know what that meant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 47 | 40 | 87
units on a scale
  Following a generally healthy diet | 0.23 (2.50) | 0.96 (2.74) | 0.57 (2.62)
  Following a disease specific diet plan | 0.29 (1.85) | 0.45 (1.85) | 0.36 (1.84)
  Self-monitoring blood glucose as advised by a h | -0.66 (3.19) | -0.18 (2.40) | -0.44 (2.84)
  Checking feet daily for wounds | -0.81 (2.64) | 0.01 (1.93) | -0.43 (2.36)
  Carb Spacing carbohydrates throughout the day: number analyzed (Participants) | 47 | 39 | 86
  Carb Spacing carbohydrates throughout the day | 0.11 (4.51) | 0.31 (3.89) | 0.20 (4.22)
  Getting sufficient physical activity | 0.11 (2.97) | 0.81 (2.88) | 0.43 (2.94)

13. Secondary Outcome: Change in Wilson 3 Item Scale From Baseline
Description: Medication adherence(Wilson et al.,2014). The 3item medication adherence scale is a self-report measure that assessing no. of days medication missed in prior month, days taken medication as advised & self-rated medication adherence. Developed in HIV research, it has been validated for non-HIV medications (Wilson, et al,2016). Each component contributes 33% of the scale. Total score ranges from 0-100. It is the combination of 3 sub-scores, (days missed dose(negative scored), self-rating, days taking medications as indicated). Higher scores indicate better medication adherence.
Time Frame: 6 Months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 52 | 46 | 98
units on a scale | -15.73 (30.87) | -12.39 (31.11) | -14.16 (30.87)

14. Secondary Outcome: Change in Wilson 3 Item Scale From 6 Months to 12 Months
Description: as for outcome 13
Time Frame: 12 Months
Population: 1 Participant decline to answer question
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 46 | 40 | 86
units on a scale | 1.74 (18.92) | 3.22 (22.89) | 2.43 (20.75)

15. Secondary Outcome: Change in Healthcare Utilization From Baseline
Description: Healthcare utilization by EMR review of clinic appointments, ED visits and hospitalizations within enrollment through 6 months at each follow up visit.
Time Frame: 6 Months
Population: 166 patients who initially enrolled followed in EMR
Measure: Mean (Standard Deviation); unit: Number of Healthcare Encounters
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 86 | 80 | 166
Number of Healthcare Encounters
  ED/UCC Visit | 1.47 (1.87) | .88 (2.22) | 1.18 (2.06)
  Hospitalization | 0.24 (.72) | .13 (.96) | .19 (.84)
  Clinic Visits Made | -.97 (3.87) | -2 (6.45) | -1.46 (5.28)

16. Secondary Outcome: Change in Healthcare Utilization From 6 Months to 12 Months
Description: as for outcome 15
Time Frame: 12 Months
Population: all patients initially enrolled in trial followed in EMR
Measure: Mean (Standard Deviation); unit: Number of Healthcare Encounters
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 86 | 80 | 166
Number of Healthcare Encounters
  ED/UCC Visit | 0.07 (1.35) | .05 (1.57) | .06 (1.46)
  Hospitalization | -.02 (.65) | 0 (.83) | -.01 (.74)
  Clinic Visits Made | 1.10 (4.30) | .88 (6.30) | .99 (5.34)

17. Secondary Outcome: Change in Diabetes Empowerment Scale Short Form From Baseline
Description: Change in Self-efficacy. Diabetes Empowerment Scale Short Form (Anderson, Fitzgerald, Gruppen, Funnell, & Oh, 2003), is a measure of a patient's overall diabetes related self-efficacy, shortened by the original from 37 to an 8 item scale. It has reliability of alpha=0.84; and has been shown to be sensitive to change in multiple populations and is correlated with improved glycemic control measured by A1C (Anderson et al., 2003). It ranges from 8-40 points; higher score indicates higher self-efficacy.
Time Frame: 6 Months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 52 | 46 | 98
units on a scale | -0.17 (0.63) | -0.05 (0.69) | -0.11 (0.66)

18. Secondary Outcome: Change in Diabetes Empowerment Scale Short Form From 6 Months to 12 Months
Description: as for outcome 17
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 47 | 40 | 87
units on a scale | 0.13 (0.49) | -0.03 (0.54) | 0.05 (0.52)

19. Secondary Outcome: Change in Diabetes Distress Scale From Baseline
Description: Diabetes related distress (Diabetes Distress Scale) (Polonsky et al., 2005), is a 17 item scale measuring distress related to emotional burden, physician-related distress, regimen-related distress, and diabetes-related interpersonal issues. It has a Cronbach's alpha of 0.88-0.93 in various studies. Higher scores are negatively correlated with several healthy behaviors. Each question is a Likert scale ranking of how serious a particular issue is from 1-6, 6 indicating a more significant problem. The scores are then averaged across all item, with final scores ranging from 1-6, with 6 indicating higher levels of distress
Time Frame: 6 Months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 52 | 46 | 98
units on a scale | 0.65 (0.97) | 0.60 (1.15) | 0.63 (1.06)

20. Secondary Outcome: Change in Diabetes Distress Scale From 6 Months to 12 Months
Description: as for outcome 19
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 47 | 40 | 87
units on a scale | 0.06 (0.92) | -0.01 (0.71) | 0.03 (0.83)

21. Secondary Outcome: Change in Patient Health Questionnaire 9 From Baseline
Description: Depression as measured by the PHQ-9 (Kroenke, Spitzer, Williams, & Lowe, 2010), is a widely used scale of depression used in clinical practice and research. The Cronbach's alpha ranges from 0.86-0.89, and it has been validated in multiple languages. Depression is worse with higher scores. Score ranges from 0 to 27. Higher levels of depression are associated with fewer healthy behaviors and worse glycemic control.
Time Frame: 6 Months
Population: 2 participants in active control arm did not attend follow up visit. Hba1c taken from medical records, no other data available. 1 participant decline to answer question
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 51 | 46 | 97
units on a scale | 3.86 (6.19) | 2.33 (6.20) | 3.13 (6.21)

22. Secondary Outcome: Change in Patient Health Questionnaire 9 From 6 Months to 12 Months
Description: as for outcome 21
Time Frame: 12 Months
Population: 2 participants decline to answer questions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 45 | 40 | 85
units on a scale | -0.18 (6.86) | -0.13 (5.17) | -0.15 (6.09)

23. Secondary Outcome: Change in Fatalism From Baseline
Description: Fatalism is measured by the Diabetes Fatalism Scale (Egede & Ellis, 2010), which measures three subscale emotional distress, religiosity and coping and perceived self-efficacy, which are summed together. The total score ranges from 12-72, higher score indicates higher fatalism, and has a Cronbach's alpha of 0.80. The score is associated with glycemic control, depression, self-care behaviors and social factors.
Time Frame: 6 Months
Population: 2 participants decline to answer questions. 2 participants in active control arm did not attend follow up visit. Hba1c taken from medical records, no other data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 50 | 46 | 96
units on a scale | -1.44 (9.47) | 0.58 (10.61) | -0.47 (10.03)

24. Secondary Outcome: Change in Fatalism From 6 Months to 12 Months
Description: as for outcome 23
Time Frame: 12 Months
Population: 5 participants decline to answer questions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 44 | 38 | 82
units on a scale | -1.30 (8.97) | -1.20 (8.51) | -1.26 (8.70)

25. Secondary Outcome: Change in WHO Quality of Life From Baseline
Description: Quality of life (World Health Organization WHO-5 Well Being Index) (Topp, Ostergaard, Sondergaard, & Bech, 2015) is a widely used measure of quality life, validated in many languages and consists of only 5 items. Each self-reported item is scored between 0 and 5, summed together and then multiplied by 4. The total range is from 0 to 100, with 0 being the lowest quality of life.
Time Frame: 6 Months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 52 | 46 | 98
units on a scale | -9.69 (31.47) | -4.96 (29.86) | -7.47 (30.66)

26. Secondary Outcome: Change in WHO Quality of Life From 6 Months to 12 Months
Description: as for outcome 25
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 47 | 40 | 87
units on a scale | 0.09 (34.02) | 6.30 (29.90) | 2.94 (32.16)

27. Secondary Outcome: Change in Diabetes Family Behavior Checklist - Supportive From Baseline
Description: Diabetes-related supportive and obstructive family behaviors are measured by patient report on the Diabetes Family Behavior checklist (Lewin et al., 2005). Family behaviors: supportive and non-supportive sub-scores of the Diabetes Family Behavior Checklist: supportive ranges from 4-45 (4 being lowest in family supportive behavior), non-supportive ranges from 7-35 (4 indicating least report of non-supportive behavior). Non-supportive scores are subtracted form supportive scores for a total.
Time Frame: 6 Months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 52 | 46 | 98
units on a scale | .58 (7.99) | .12 (9.08) | .36 (8.48)

28. Secondary Outcome: Change in Diabetes Family Behavior Checklist Supportive From 6 Months to 12 Months
Description: as for outcome 27
Time Frame: 12 Months
Population: patients who achieved follow up at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 47 | 40 | 87
units on a scale | -.70 (7.87) | -.98 (9.32) | -.83 (8.52)

29. Secondary Outcome: Change in Diabetes Family Behavior Checklist - Nonsupportive From Baseline
Description: as for outcome 27
Time Frame: 6 Months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 52 | 46 | 98
units on a scale | .58 (6.25) | .56 (6.86) | .57 (6.51)

30. Secondary Outcome: Change in Diabetes Family Behavior Checklist Nonsupportive From 6 Months to 12 Months
Description: as for outcome 27
Time Frame: 12 Months
Population: patients who achieved follow up at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 47 | 40 | 87
units on a scale | -.85 (6.10) | -1.13 (6.93) | -.98 (6.46)

31. Secondary Outcome: Change in Diabetes Care Profile Support From Baseline
Description: Diabetes-specific social support is measured by the Diabetes Care Profile Support Questions,(Fitzgerald et al., 1996) with sub-scores for perceived disease specific support needs and perceived disease specific support received. Diabetes Care Profile support questions: Support wanted, and support received. Each range from 5 to 30, high scores indicating high desire for support and higher support received.
Time Frame: 6 Months
Population: as for outcome 11
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 52 | 46 | 98
units on a scale
  Perceived Disease Specific Support Needs | 4.44 (10.79) | 5.80 (9.06) | 5.08 (9.99)
  Perceived Disease Specific Support Received | -0.08 (9.68) | -3.65 (9.11) | -1.76 (9.54)
  Support Attitudes | 0.96 (6.51) | -0.87 (5.73) | 0.10 (6.20)

32. Secondary Outcome: Change in Diabetes Care Profile Support From 6 Months to 12 Months
Description: as for outcome 31
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 47 | 40 | 87
units on a scale
  Perceived Disease Specific Support Needs | -0.38 (8.17) | 0.40 (10.31) | -0.02 (9.17)
  Perceived Disease Specific Support Received | -1.38 (7.54) | 2.70 (8.17) | 0.49 (8.06)
  Support Attitudes | -0.77 (4.56) | 0.08 (4.01) | -0.38 (4.31)

33. Secondary Outcome: Change in Norbeck Social Support Questionnaire From Baseline
Description: Measure Description: General social support is captured by the Norbeck Social Support Questionnaire Emotional and&Tangible subscales.(Norbeck, Lindsey, & Carrieri, 1981) General social support: Norbeck Social Support Questionnaire, emotional sub score (ranges 0-16, with higher scores indicating higher perceived emotional support) & tangible sub score (0-8, higher score indicating higher perceived tangible support). While the subscores are highly correlated, the authors do not recommend Cronbach's alpha as a test of internal validity.(http://eileengigliotti.com/uploads/1/1/0/2/110241155/nssq-psychometric.pdf)
Time Frame: 6 Months
Population: 10 participants decline to answer questions. 2 participants in active control arm did not attend follow up visit. Hba1c taken from medical records, no other data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 47 | 41 | 88
units on a scale
  Emotional | 0.64 (4.02) | -0.22 (4.41) | 0.24 (4.20)
  Tangible | 0.06 (1.99) | -0.29 (2.02) | -0.10 (2.00)

34. Secondary Outcome: Change in Norbeck Social Support Questionnaire From 6 Months to 12 Months
Description: as for outcome 33
Time Frame: 12 Months
Population: 2 participants decline to answer question
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 46 | 39 | 85
units on a scale
  Emotional | -0.48 (4.03) | 0.69 (4.01) | 0.06 (4.04)
  Tangible | -0.36 (2.17) | 0.48 (2.08) | 0.02 (2.16)

35. Secondary Outcome: Change in Partner Distress Scale From Baseline
Description: Supporter diabetes-related distress is measured by the Partner Distress Scale (Polonsky, Fisher, Hessler, &Johnson, 2016). The self-report scale consists of 21 items in 4 domains: "my partner's diabetes management", "how best to help", "diabetes & me", & "hypoglycemia". Domains are summed together. Each item is score from 0 to 4, lower scores indicate less distress. The total score is an average of the 21 items. The Cronbach's alpha was 0.76 for total scores. Greater partner distress is correlated with higher A1C among patients, worse self-care & lower satisfaction with relationship
Time Frame: 6 Months
Population: Supporters who were reached for follow up at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED+FANS | Total
Number analyzed (Participants) | 62 | 54 | 116
units on a scale | .45 (0.83) | .13 (.89) | .37 (.89)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | TExT-MED Only | TExT-MED+FANS
All-Cause Mortality (participants affected / at risk) | 0/86 | 1/80
Serious Adverse Events (participants affected / at risk) | 21/86 | 19/80
Other Adverse Events (participants affected / at risk) | 0/86 | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TExT-MED Only (N=86) | TExT-MED+FANS (N=80)
Report of Hypoglycemic events (Endocrine disorders) | 21 (32) | 19 (24) — Patient reporting a subjective or measured hypoglycemic event

LIMITATIONS AND CAVEATS:
Follow up rates were lower than anticipated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT03178773/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT03178773/SAP_001.pdf
  • Informed Consent Form (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT03178773/ICF_002.pdf